CLINICAL TRIAL: NCT03255031
Title: Ketogenic Diet (KD) in Alcoholism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 170152; 17-AA-0152
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-01-25

CONDITIONS: Alcoholism
Keywords: Ketogenic Diet; Detoxification; Functional MRI; MRI/MRS; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Diet, Ketogenic; Meals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (KD) (Active Comparator): Subjects with alcohol use disorder receive ketogenic diet (KD) which consists of food, snacks, and shakes three times per day (high in fat) for up to four weeks while inpatient.
  Interventions: Other: Ketogenic Diet (KD)
- Standard American (SA) diet (Placebo Comparator): Subjects with alcohol use disorder receive Standard American (SA) diet which consists of ketogenic diet (KD) food, snacks, and shakes three times per day (high in fat) in the proportions of carbohydrates, protein and fat of traditional western diet for up to four weeks while inpatient.
  Interventions: Other: Standard American (SA) Meals and Shakes

INTERVENTIONS:
Other: Ketogenic Diet (KD) — For each meal at breakfast, lunch and dinner, the diets will consist of ketogenic diet (KD) meal. Compliance tests are done twice a week with a blood test measuring ketone levels.
  Arms: Ketogenic diet (KD)
Other: Standard American (SA) Meals and Shakes — For each meal at breakfast, lunch and dinner, the diets will consist of SA meal (carbohydrate rich) KD meal. Compliance tests are done twice a week with a blood test measuring ketone levels.
  Arms: Standard American (SA) diet

SUMMARY:
Background:

A ketogenic diet (KD) is high in fat and low in carbohydrates. Research has shown that a KD can lessen tremor in animals withdrawing from alcohol. KD can also help people who have difficulties with thinking, sleep, and mood. Researchers want to see if KD can lessen symptoms of alcohol withdrawal in people with alcohol use disorder.

Objective:

To test the effects of a ketogenic diet on alcohol withdrawal symptoms.

Eligibility:

Adults 18 years or older who are moderate or severe alcohol drinkers and are seeking treatment for alcohol use. They must be in the NIAAA inpatient alcohol treatment program.

Design:

Participants will be screened under another protocol. They will have a medical and psychiatric history, physical exam, and blood and urine tests. Participants will have a breath test for alcohol.

The study will be done in a 3-week stay in the clinic.

Participants will get either a KD or Standard American diet.

Participants will have breathalyzer, blood, and urine tests.

Participants will have magnetic resonance imaging (MRI) scans. The scanner is a cylinder in a magnetic field. They will lie on a table that slides in and out of the cylinder. They will do tasks on a computer during the scan.

Participants will have tests of thinking, memory, and attention.

Participants will have their sleeping and waking measured. They will wear a device like a headband held in place with elastic straps. Several electrodes will be placed on the body.

Participants will have heart tests.

Participants will wear an activity monitor on the wrist.

After the clinic stay, participants will be called by phone about 5 times over 3 months.

DETAILED DESCRIPTION:
Alcohol intoxication leads to marked reductions in brain glucose metabolism that reflect in part the use of ketones (including acetate) as alternative energy sources by the brain during intoxication. With repeated alcohol exposure both clinical and preclinical studies have shown a shift of brain substrate preference towards ketones. This has led us to question the potential value of a ketogenic diet in alcohol detoxification in order to prevent the ketone deprivation that would follow alcohol detoxification in alcoholics.

Objectives: Here we propose a blinded randomized design to assess the effects of a ketogenic diet on symptoms of alcohol withdrawal and on brain function in alcoholics undergoing inpatient treatment of alcohol detoxification. We hypothesize that a ketogenic diet will increase acetate levels in brain resulting in improved brain function in alcoholics as well as a reduction of alcohol withdrawal symptoms during detoxification.

Study population: Participants diagnosed with alcohol use disorder (AUD) as per Diagnostic and Statistical Manual (DSM) IV or DSM 5. Males and females ages 18 years and older will be included.

Design: This will include an inpatient component and outpatient follow-up. Patients are admitted to the Clinical Center (CC) for detoxification, where they undergo treatment as usual (TAU) and will be randomized into a regular versus a ketogenic diet. Patients will be given benzodiazepines only if withdrawal symptoms emerge while receiving either the ketogenic or the regular diet. Within 2-6 days after admission, all patients will undergo an MRI (brain structure and function, functional connectivity and spectroscopy, i.e. MRS) and a battery of neuropsychological tests (NP). MRI scans will also be obtained in week 2. After 3 weeks of inpatient care the MRI scans and NP studies will be repeated. We will complete all study procedures in n=25 patients with AUD with the ketogenic diet and n=25 with the regular diet.

Outcome parameters: Main outcome: To assess the effects of a ketogenic diet in patients hospitalized for the treatment of alcohol detoxification, on: (1) withdrawal symptoms including the need of medications to control them (benzodiazepines); (2) brain function as assessed by functional magnetic resonance imaging (fMRI) (at rest and during task conditions), (3) MRS, and (4) structural MRI. Secondary Outcomes: To assess the effects of a ketogenic diet on performance of cognitive tests, sleep, mood and craving.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with AUD

1. Age 18 years and older.
2. Ability to provide written informed consent as determined by clinical examination and verbal communication. Capacity to consent will be determined by those giving the informed consent.
3. DSM-IV diagnosis of alcohol dependence or alcohol abuse or DSM 5 diagnosis of moderate or severe AUD (established through history and clinical exam).
4. Participants seeking treatment for their AUD (self-report)
5. Minimum 5-year history of heavy drinking (SAMSHA s criteria for heavy drinking: for men 5 or more drinks/day on at least 5 different days per month; and for women 4 or more drinks/day on at least 5 different days per month [self-report]).
6. Alcohol specified as the preferred drug (self-report).
7. NIH employees with an AUD may participate in this study.

EXCLUSION CRITERIA:

1. Unwilling or unable to refrain from use, within 24 hours of MRI and NPT procedures, psychoactive medications or medication that may affect study results (e.g., analgesics containing narcotics, antibiotics [must finish course at least 24 hours prior to a scheduled procedure], antidiarrheal preparations, anti-inflammatory drugs [systemic corticosteroids are exclusionary], antinauseants, cough/cold preparations) (self-report, medical history). The following medications are allowable for entry on this study: analgesics (non-narcotic); antacids; antiasthma agents that are not systemic corticosteroids; antifungal agents for topical use; antihistamines (non-sedating); H2-Blockers/proton pump inhibitors (PPI); laxatives. The use of antihyperlipidemics and/or diuretics are permitted as long as they have been taken for at least 1 month before procedure visits and dose has been stabilized.
2. Current DSM-IV or DSM 5 diagnosis of a major psychiatric disorder (other than alcohol and nicotine use disorders, or substance use disorders that are mild/moderate) that required hospitalization, or that required daily medications for over 4 weeks in the past year (i.e., antidepressants; anticholinergics; antipsychotics; anxiolytics; lithium; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics). Chronic benzodiazepine use prior to alcohol detox will also be excluded. Note that nicotine and/or caffeine use will not exclude participation.
3. Chronic use of the following medications: analgesics containing narcotics; anorexics (sibutramine); antianginal agents; antiarrhythmics; antiasthma agents that are systemic corticosteroids; antibiotics; anticoagulants; anticonvulsants; antidiarrheal preparations; antifungal agents (systemic); antihistamines (sedating); antihypertensives (except angiotensin - converting

   enzyme (ACE) inhibitors such as Lisinopril, or Angiotensin receptor blockers (ARB) such as Losartan); anti-inflammatory drugs (systemic); antineoplastics; antiobesity; antivirals (except for treatment of HSV with agents without CNS activity, e.g. acyclovir, ganciclovir, famciclovir, valacyclovir); cough/cold preparations (dextromethorphan preparations, pseudoephedrine); hormones (exceptions: thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy); insulin; and muscle relaxants.
4. Major medical problems that can impact brain function or the use of a ketogenic diet (e.g., epilepsy, diabetes, liver disease, kidney disease, kidney stones (current and/or in the past), chronic metabolic acidosis or a cardiomyopathy) as determined by EKG, history and clinical exam.
5. Clinically significant laboratory findings that could affect brain function (e.g. HIV+).
6. Head trauma with loss of consciousness for more than 30 minutes (self-report, medical history).
7. Pregnant or breast-feeding: Females of childbearing potential, or with tubal ligation, or are post-menopausal and are age 60 or less will undergo a urine pregnancy test and it must be negative to continue participation. Urine pregnancy tests will be repeated on subsequent days of study. (i.e., within 24 hours before study procedures). Females must not be currently breastfeeding.
8. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head, fear of enclosed spaces, or other standard contraindication to MRI (self-report checklist).
9. Cannot lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
10. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 0 lbs.
11. Milk or soy allergy (self-report).

Note that subjects will not be excluded on initial screening from enrollment onto this study if their breath alcohol test is positive; or if their urine test is positive for drugs. The following guideline will be followed for positive alcohol/drug screens on study procedure days:

-If an AUD subject s breath alcohol and/or urine drug screen test is/are positive on study days (i.e., within 24 hours before study procedures except for benzodiazepines during detox, including oxazepam [Serax], the procedures will be postponed and rescheduled to another day. If the urine drug screen is positive for THCCOOH, a saliva drug screen will be performed and subject may proceed with MRI/NPT procedures if saliva results for Delta-9-Tetrahydrocannabinol (THC) are negative. We will not place a limit on rescheduling study days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene-Jack Wang, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.Data is analyzed by subject group and not on an individual basis.

REFERENCES:
- [Result] Wiers CE, Vendruscolo LF, van der Veen JW, Manza P, Shokri-Kojori E, Kroll DS, Feldman DE, McPherson KL, Biesecker CL, Zhang R, Herman K, Elvig SK, Vendruscolo JCM, Turner SA, Yang S, Schwandt M, Tomasi D, Cervenka MC, Fink-Jensen A, Benveniste H, Diazgranados N, Wang GJ, Koob GF, Volkow ND. Ketogenic diet reduces alcohol withdrawal symptoms in humans and alcohol intake in rodents. Sci Adv. 2021 Apr 9;7(15):eabf6780. doi: 10.1126/sciadv.abf6780. Print 2021 Apr. PMID 33837086
- [Result] Li X, Shi Z, Byanyima J, Morgan PT, van der Veen JW, Zhang R, Deneke E, Wang GJ, Volkow ND, Wiers CE. Brain glutamate and sleep efficiency associations following a ketogenic diet intervention in individuals with Alcohol Use Disorder. Drug Alcohol Depend Rep. 2022 Dec;5:100092. doi: 10.1016/j.dadr.2022.100092. Epub 2022 Sep 8. PMID 36311277
- [Result] Wiers CE, Manza P, Wang GJ, Volkow ND. Ketogenic diet reduces a neurobiological craving signature in inpatients with alcohol use disorder. Front Nutr. 2024 Feb 12;11:1254341. doi: 10.3389/fnut.2024.1254341. eCollection 2024. PMID 38410637
- [Derived] Zhang R, Tomasi D, Shokri-Kojori E, Manza P, Feldman DE, Kroll DS, Biesecker CL, McPherson KL, Schwandt M, Wang GJ, Wiers CE, Volkow ND. Effect of detoxification on N3 sleep correlates with brain functional but not structural changes in alcohol use disorder. Drug Alcohol Depend. 2022 Sep 1;238:109545. doi: 10.1016/j.drugalcdep.2022.109545. Epub 2022 Jun 26. PMID 35779511
- [Derived] Bornebusch AB, Mason GF, Tonetto S, Damsgaard J, Gjedde A, Fink-Jensen A, Thomsen M. Effects of ketogenic diet and ketone monoester supplement on acute alcohol withdrawal symptoms in male mice. Psychopharmacology (Berl). 2021 Mar;238(3):833-844. doi: 10.1007/s00213-020-05735-1. Epub 2021 Jan 7. PMID 33410985
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-AA-0152.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Started | 33 | 20
Completed | 17 | 13
Not Completed | 16 | 7
Not completed — Adverse Event | 5 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet | Total
Number analyzed (Participants) | 33 | 20 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 18 | 51
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 21 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 30 | 17 | 47
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 16 | 8 | 24
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 20 | 53

OUTCOME MEASURES:

1. Primary Outcome: Withdrawal Symptoms Measured Using the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar)
Description: Alcohol withdrawal symptoms were measured using the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar). The CIWA-Ar is a 10-item scale scored from 0-7, with the exception of the orientation category, scored from 0-4, used in the assessment and management of alcohol withdrawal. Score ranges from 0 - 67. Mild alcohol withdrawal is defined with a score less than or equal to 10, moderate with scores 11 to 15, and severe with any score equal to or greater than 16. Analysis was performed as ANOVA between-groups.
Time Frame: Week 1
Population: The analyses included participants who completed the dietary intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
score on a scale | 4.16 (3.962) | 6.57 (5.345)
Statistical Analysis 1: Comparison: Ketogenic Diet (KD) vs Standard American (SA) Diet; Test type: Superiority; p = 0.067, Mixed Models Analysis — The threshold for statistical significance was p = 0.05

2. Primary Outcome: Quantification of Medications for Control of Withdrawal Symptoms
Description: Participants received oral benzodiazepine treatment for alcohol withdrawal when Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) scores were 8 or higher within the first week of inpatient admission. The effect of alcohol withdrawal and benzodiazepine use was analyzed with ANOVA as the group × time effect on benzodiazepine use.
Time Frame: Week 1
Population: The analyses included participants who completed the dietary intervention.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
mg | 34.21 (79.395) | 156.43 (206.234)
Statistical Analysis 1: Comparison: Ketogenic Diet (KD) vs Standard American (SA) Diet; Test type: Superiority; p = 0.004, Mixed Models Analysis — The threshold for statistical significance was p = 0.05

3. Primary Outcome: Brain Functions During Resting State: Sensorimotor Brain Network
Description: Brain network segregation was measured by functional MRI (fMRI) using the Power-264 brain atlas. The 264 spherical is defined as brain regions of interest (ROIs) with a 5-mm radius that belong to 13 large-scale functional brain networks. The fronto-parietal, ventral attention, dorsal attention, cingulo-opercular, and salience networks were grouped into the association network. The sensory hand, sensory mouth, visual, and auditory networks were grouped into the sensorimotor network. The mean time series across voxels was extracted for each regions of interest. Then the Pearson correlation coefficients was calculated between the ROIs and converted to Fisher-Z values for further analysis. Segregation equals the relative strength of within-network connectivity (Zw) when compared with between-network connectivity (Zb): Zw - Zb / Zw. Higher segregation value corelates with better functional specificity and energy efficiency. The final segregation output is a ratio of Z-scores.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and had fMRI testing.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 17 | 13
Ratio
  Week 1 | 0.5314 (0.0681) | 0.4816 (0.0844)
  Week 2 | 0.5067 (0.0496) | 0.5028 (0.3346)
  Week 3 | 0.4932 (0.0671) | 0.4849 (0.0749)

4. Primary Outcome: Brain Functions During Resting State: Association Brain Network
Description: Brain network segregation was measured by functional MRI (fMRI) using the Power-264 brain atlas. The 264 spherical is defined as brain regions of interest (ROIs) with a 5-mm radius that belong to 13 large-scale functional brain networks. The fronto-parietal, ventral attention, dorsal attention, cingulo-opercular, and salience networks were grouped into the association network. The sensory hand, sensory mouth, visual, and auditory networks were grouped into the sensorimotor network. The mean time series across voxels was extracted for each regions of interest. Then the Pearson correlation coefficients was calculated between the ROIs and converted to Fisher-z values for further analysis. Segregation equals relative strength of within-network connectivity when compared with between-network connectivity: Zw - Zb / Zw. Higher segregation value corelates with better functional specificity and energy efficiency. The final segregation output is a ratio of Z-scores.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and had fMRI testing.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 17 | 13
Ratio
  Week 1 | 0.3647 (0.0537) | 0.3125 (0.0591)
  Week 2 | 0.3624 (0.0445) | 0.3346 (0.0734)
  Week 3 | 0.3563 (0.0574) | 0.3206 (0.06657)

5. Primary Outcome: Neurobiological Craving Signature (NCS) for Alcohol > Food Pictorial Cues
Description: Participants performed an alcohol cue-reactivity paradigm with functional magnetic resonance imaging in which they viewed alcohol and food pictorial cues. The blood-oxygen-level dependent (BOLD) responses to food and alcohol cues was extracted and quantified the degree to which each set of brain images shared a pattern of activation using the Neurobiological Craving Signature (NCS). The NCS is a whole-brain pattern of responses to cues, with prominent regions including ventromedial prefrontal and cingulate cortices, ventral striatum, temporal/parietal association areas, mediodorsal thalamus and cerebellum. A group-by-time repeated measures ANOVA was used to test for differences in craving signature expression between the dietary groups. Positive values indicate stronger brain BOLD responses to alcohol related cues.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and the fMRI tests.
Measure: Mean (Standard Deviation); unit: arbitrary units (A.U)
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
arbitrary units (A.U)
  Week 1 | -2.13 (3.6952873396632) | .55 (4.2818982698951)
  Week 2 | -2.38 (4.2621609031125) | -.67 (3.5104963867952)
  Week 3 | -1.37 (3.2654308575651) | -.099 (5.8017946230225)

6. Primary Outcome: Brain Concentrations of Glutamate/Creatine
Description: The brain metabolism was measured with weekly magnetic resonance spectroscopy (MRS) scans in a voxel in the dorsal anterior cingulate cortex. The concentrations of Glutamate/Creatine were analyzed with repeated-measures ANOVAs with time as the within-subject factor and diet as the between-subject factor.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and the MRS exam.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
Ratio
  Week 1 | 1.1980558 (.13154360) | 1.1966429 (.15106015)
  Week 2 | 1.34895 (.214281) | 1.20654 (.103377)
  Week 3 | 1.31244 (.169988) | 1.18600 (.164481)

7. Primary Outcome: Brain Volume Measured With Brain MRI
Description: Whole brain total intracranial volume was measured using T1 structural MRI. Voxel-based morphometry (VBM) was performed using the Computational Anatomy Toolbox (CAT12) in Statistical Parametric Mapping software (SPM12).
Time Frame: Weeks 1 and 3
Population: The analyses included participants who completed the dietary intervention and MRI exams.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 18 | 12
cm^3
  Week 1 | 1482.111 (158.8806) | 1462.667 (143.786)
  Week 3 | 1481.0 (161.053) | 1463.75 (147.00)

8. Secondary Outcome: Effect of Ketogenic Diet on Mood
Description: The effect of ketogenic diet on mood was assessed with the Montgomery-Asberg Depression Rating Scale (MADRS). MADRS is a ten-item diagnostic questionnaire which measures the severity of depressive episodes. Each item is rated on a score of 0 (normal/not present) to 6 (extreme symptom). Total score range is zero (0) to 60. Total score of 7-19 represent mild depression; 20-34 moderate; 35-60 indicate severe depression. Higher MADRS score indicates more severe depression/lower mood. Analysis was performed as mixed ANOVAs with group as between-group factor and time as within-subjects factor.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and the MADRS scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
score on a scale
  Week 1 | 18.22 (8.968) | 21.71 (12.086)
  Week 2 | 6.39 (7.632) | 7.29 (3.872)
  Week 3 | 6.26 (6.297) | 6.36 (6.902)

9. Secondary Outcome: Effect of Ketogenic Diet on Sleep
Description: Participants self-reported their estimated total sleep time for each night. Weekly responses were reported as the average across seven days.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and reported sleep data.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
Hours
  Week 1 | 5.6451754385263 (1.0673525108302) | 6.0624149660000 (1.0478988048910)
  Week 2: number analyzed (Participants) | 19 | 13
  Week 2 | 5.7086466163684 (.75371098816986) | 6.1456632652857 (1.0118081840508)
  Week 3 | 5.6344611528421 (.87434796211452) | 6.5103741495714 (.78393883493517)

10. Secondary Outcome: Effect of Ketogenic Diet on Alcohol Craving
Description: Participants rated their alcohol craving on the Desire for Alcohol Questionnaire (DAQ) weekly. DAQ is a 14-item scale that assesses current self-reported levels of alcohol craving. Each item is scored from 0 (fully disagree) to 6 (fully agree), with a total score range of zero (0) to maximum score of 84. Higher score indicates higher level of alcohol craving. Analysis was performed as repeated-measure ANOVA.
Time Frame: Weeks 1, 2, and 3
Population: The analyses included participants who completed the dietary intervention and completed the DAQ. Two participants from week 3 had missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
Number analyzed (Participants) | 19 | 14
score on a scale
  Week 1 | 22.00 (16.327) | 21.07 (16.041)
  Week 2 | 17.53 (11.649) | 20.36 (16.402)
  Week 3: number analyzed (Participants) | 17 | 14
  Week 3 | 15.88 (10.511) | 18.36 (11.098)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks while inpatient
Arm/Group | Ketogenic Diet (KD) | Standard American (SA) Diet
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/20
Other Adverse Events (participants affected / at risk) | 5/33 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketogenic Diet (KD) (N=33) | Standard American (SA) Diet (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Liver function test increased (Investigations) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03255031/Prot_SAP_000.pdf